CLINICAL TRIAL: NCT06708299
Title: IMpAct of CardiolRxTM oVer 6 Months Following IL-1 Blocker Cessation in pERICarditis Patients - MAVERIC A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: CardiolRx in Recurrent Pericarditis Following IL-1 Blocker Cessation
Acronym: MAVERIC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cardiol Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Cardiol 100-006
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Pericarditis
Keywords: IL-1 blocker-dependent recurrent pericarditis; pharmaceutically cannabidial
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CardiolRx (Active Comparator): * Initial starting dose (Day 1, evening dose to Day 3, morning dose):
    5 mg/kg of body weight CardiolRx b.i.d.
  * Day 3, evening dose to Day 10, morning dose: 7.5 mg/kg of body weight CardiolRx b.i.d.
  * Day 10, evening dose to morning dose of the Week 24 Visit:
    10 mg/kg of body weight CardiolRx b.i.d.
  Interventions: Drug: CardiolRx
- Placebo (Placebo Comparator): * Initial starting dose (Day 1, evening dose to Day 3, morning dose):
    5 mg/kg of body weight matching placebo b.i.d.
  * Day 3, evening dose to Day 10, morning dose: 7.5 mg/kg of body weight matching placebo b.i.d.
  * Day 10, evening dose to morning dose of the Week 24 Visit:
    10 mg/kg of body weight matching placebo b.i.d.
  Interventions: Drug: CardiolRx

INTERVENTIONS:
Drug: CardiolRx — The intervention will be administered orally (via syringe) with food twice daily.
  Other Names: Pharmaceutically produced cannabidiol

SUMMARY:
Multi-center, randomized, double-blind, placebo-controlled, phase-3 Trial. Patients with a history of recurrent pericarditis who are being treated with an IL-1 blocker for at least 12 months, scheduled to be discontinued, will be approached for potential trial participation.

Double-blind treatment will be initiated 10 - 16 days prior to the last scheduled dose of the IL-1 blocker and continued for 24 weeks.

The objective is to assess whether patients who discontinue therapy with an IL-1 blocker for recurrent pericarditis remain free of pericarditis recurrence while receiving CardiolRx.

DETAILED DESCRIPTION:
Double-blind, randomized, placebo-controlled Phase-3 trial. The primary objective is to assess whether patients with IL-1 blocker-dependent recurrent pericarditis can discontinue IL-1 blocker therapy and remain free of recurrence while receiving CardiolRx.

Before any trial-related procedure is performed, written informed consent will be obtained. After informed consent is obtained, patients will be screened for eligibility.

The highest NRS pain score within the past 7 days is to be assessed prior to randomization at Visit 1 (Day 1). Baseline blood samples for central laboratory assessment of hs-CRP and pharmacokinetic assessments should also be collected prior to randomization at Visit 1 (Day 1).

All other screening assessments will be performed at any time within 7 days prior to randomization at Visit 1 (Day 1) and include the following: Physical examination, vital signs, 12-lead ECG; C-SSRS and blood draws for local laboratory assessments (see Section 17.2).

Eligible patients will be randomized at Visit 1 (Day 1) to either CardiolRx or matching placebo in a 1:1 ratio. Double-blind trial therapy will be initiated in the evening of Day 1, 10 - 16 days (no additional time window is allowed) prior to the last scheduled dose of the IL-1 blocker and after all baseline assessments are completed. Trial therapy will be administered for 24 weeks.

Vital signs, ECG recording and blood draws for local and central laboratory analyses will be carried out at selected visits. Concomitant medications and (S)AEs will be recorded at all visits.

Final efficacy assessments will take place at Visit 9, 24 weeks after randomization and start of trial therapy and include a physical exam, vital signs, pain score NRS collection, a 12-lead ECG, a C-SSRS, as well as blood draws for local and central laboratory assessments.

A virtual safety follow-up visit (Visit 10) will be scheduled 4 weeks after the last trial therapy administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. A history of recurrent pericarditis with stable disease and currently being treated with an IL-1 blocker, scheduled to be discontinued. Stable disease is defined as:

   * treatment with an IL-1 blocker for at least 12 months,
   * free of pericarditis recurrence for at least 6 months and this recurrence, if present, must have occurred in the setting of an interruption or tapering of an IL-1 blocker; and
   * treatment with an unchanged dose and regimen of on an IL-1 blocker for at least 3 months prior to randomization.
3. Pericarditis pain les or equal than 2 on the 11-point Numerical Rating Scale (NRS) for at least 7 days prior to randomization (Visit 1, Day 1)
4. C-Reactive Protein (CRP) < 1.0 mg/dL during screening within 7 days prior to randomization (Visit 1, Day 1).
5. Patients who have had a vasectomy or who are willing to use double barrier contraception methods with partners of childbearing potential during the conduct of the trial and for 2 months after the last dose of trial therapy.
6. Patients of childbearing potential willing to use an acceptable method of contraception starting with trial therapy administration and for a minimum of 2 months after trial completion. Otherwise, these patients must be postmenopausal (at least 1 year absence of vaginal bleeding or spotting and confirmed by follicle stimulating hormone [FSH] ≥ 40 mIU/mL [or ≥ 40 IU/L] if less than 2 years postmenopausal) or be surgically sterile.

Acceptable birth control methods that result in a failure rate of less than 1 % include oral, intravaginal or transdermal combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation; oral, injectable or implantable progestogen-only hormonal contraception associated with inhibition of ovulation; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); using double-barrier contraception methods with their partners; bilateral tubal occlusion; vasectomised partner; sexual abstinence.

Exclusion Criteria:

1. Pericarditis recurrence(s) during IL-1 blocker treatment without interruption or tapering of the IL-1 blocker
2. Diagnosis of pericarditis that is secondary to specific prohibited etiologies, including tuberculosis (TB); neoplastic, purulent, or radiation etiologies; post-thoracic blunt trauma (e.g., motor vehicle accident); systemic autoimmune disease (e.g., systemic lupus erythematosus)
3. Primary diagnosis of myocarditis (diagnosis of myopericarditis is accepted)
4. Estimated glomerular filtration rate (eGFR) < 30 mL/min during screening within 7 days prior to randomization (Visit 1, Day 1)
5. Elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limit of normal (ULN) or ALT or AST > 3x ULN plus bilirubin > 2x ULN during screening within 7 days prior to randomization (Visit 1, Day 1).
6. Sepsis, defined as documented bacteremia during screening within 7 days prior to randomization (Visit 1, Day 1) or other untreated or uncontrolled bacterial infection*
7. Prior history of sustained ventricular arrhythmia(s)
8. History of diagnosed long QT syndrome
9. QTc interval > 480 msec (biologically female) or > 470 msec (biologically male) (please refer to Section 9.2.3 for bundle branch block, bifascicular block and paced rhythm correction) or second or third degree atrioventricular (AV) block in a patient without an implanted functioning pacemaker device during screening within 7 days prior to randomization (Visit 1, Day 1)
10. Showing suicidal tendency during the last 12 months, as defined by answering "yes" to question 4 or 5 of the Columbia Suicide Severity Rating Scale (C-SSRS), administered during screening within 7 days prior to randomization (Visit 1, Day 1)
11. Participation in a clinical trial in which an investigational drug or device was administered within 30 days of screening or within 5 half-lives of the previous study drug, whichever is longer
12. Inability or unwillingness to give informed consent
13. Ongoing drug or alcohol abuse in the opinion of the investigator
14. On any cannabinoid during the past month or unwilling to stay abstinent from all cannabis products for the duration of the trial
15. Pregnant or breastfeeding
16. Current diagnosis of active cancer, with the exception of non-melanoma skin cancer
17. Any factor, which would make it unlikely that the patient can comply with the trial procedures
18. Moderate (Child-Pugh B) or severe (Child-Pugh C) hepatic impairment
19. Has received systemic immunomodulatory agents as below prior to randomization:

    1. Methotrexate (within 2 weeks)
    2. Azathioprine, mycophenolate mofetil, cyclosporine, tacrolimus, sirolimus, or mercaptopurine (within 24 weeks)
    3. Canakinumab, TNF inhibitors, IL-6 inhibitors, or janus-activating kinase inhibitors (within 12 weeks)
    4. Intravenous immune globulin (IVIG) (within 8 weeks)
    5. Corticosteroids (within 4 weeks)
20. Known hypersensitivity to the active substance or any of the excipients of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-09-21 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
Recurrence of pericarditis | 24 weeks
  proportions of patients free from a new episode of recurrent pericarditis* from the timepoint of stopping the IL-1 blocker to Week 24

SECONDARY OUTCOMES:
Percentage of days with no or minimal pain | 24 weeks
  the percentage of days with no or minimal pain as assessed by an NRS score ≤ 2 from the timepoint of stopping the IL-1 blocker to Visit 9 (Week 24)

OTHER OUTCOMES:
restricted mean time to a new episode of pericarditis recurrence | week 24
  the restricted mean time to a new episode of pericarditis recurrence from the timepoint of stopping the IL-1 blocker to Visit 9 (Week 24)
the mean pain score | week 8, week 24
  - the mean pain score using an 11-point NRS at Visit 6 (Week 8) and at Visit 9 (Week 24) (highest pain score recorded during the 7 days prior to Visit 6 and Visit 9)
the change in CRP | week 8, week 24
  - the change in CRP from Visit 1 (Day 1) to Visit 6 (Week 8) and Visit 9 (Week 24)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cremer, MD, Principal Investigator — Northwestern University
Locations (25):
- United States (19):
  - Mayo Clionic Arizona, Phoenix, Arizona
  - UCI Health, Irvine, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - MedStar Health Institute, Columbia, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Columbia University - New York Presbyterian, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Jewish General Hospital, Montreal, Canada
- Hippokration General Hospital, Athens, Greece
- Italy (4):
  - Fatebenefratelli Hospital Milano, Milan
  - University of Padua, Padua
  - University Hospital, Torino
  - University Hospital Udine, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Imazio M, Klein AL, Brucato A, Abbate A, Arad M, Cremer PC, Insalaco A, LeWinter MM, Lewis BS, Lin D, Luis SA, Nicholls SJ, Sutej P, Wasserstrum Y, Clair J, Agarwal I, Wang S, Paolini JF; RHAPSODY Investigators. Sustained Pericarditis Recurrence Risk Reduction With Long-Term Rilonacept. J Am Heart Assoc. 2024 Mar 19;13(6):e032516. doi: 10.1161/JAHA.123.032516. Epub 2024 Mar 12. PMID 38471825
- [Background] M Imazio, L Trotta, E Bizzi, M Pancrazi, S Wang, J Clair, A L Klein, E Tombetti, A Brucato, J F Paolini, RHAPSODY Investigators, Multi-year recurrent pericarditis disease duration in Italian patients: clinical outcomes after cessation of long-term IL-1 pathway inhibition provide insights for chronic management, European Heart Journal, Volume 45, Issue Supplement_1, October 2024, ehae666.2104, https://doi.org/10.1093/eurheartj/ehae666.2104